CLINICAL TRIAL: NCT04278391
Title: A Randomized, Open Label, Single Dose, Crossover Study to Compare the Pharmacokinetics and Safety Between "DWJ1421" and "DWC201903" in Healthy Male Volunteers
Brief Title: Pharmacokinetics and Safety Between "DWJ1421" and "DWC201903" in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daewoong Pharmaceutical Co. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: DW_DWJ1421101
Record Dates: First submitted 2020-02-18; First posted 2020-02-20 (Actual); Last update posted 2020-02-20 (Actual); Status verified 2020-02

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A (RT) (Experimental): Period 1 : Reference drug (DWC201903) Period 2 : Test durg(DWJ1421)
  Interventions: Drug: DWC201903
- B (TR) (Experimental): Period 1 : Test durg(DWJ1421) Period 2 : Reference drug (DWC201903)
  Interventions: Drug: DWJ1421

INTERVENTIONS:
Drug: DWJ1421 — 1 tablet administered in fasting condition
  Arms: B (TR)
Drug: DWC201903 — 1 tablet administered in fasting condition
  Arms: A (RT)

SUMMARY:
This is a randomized, open label, single dose, crossover study to compare the pharmacokinetics and safety between "DWJ1421" and "DWC201903" in healthy male volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Between 19 aged and 45 aged in healthy male adult
* Body weight more than 50kg
* Body Mass Index more than 18.0 and under 27.0

Exclusion Criteria:

* Those who have clinical significant liver, kidney, digestive system, respiratory, endocrine, nervous system, hematology and oncology, cardiovascular, urinary diseae or past history
* Those who have a gastrointestinal disease history that can effect drug absorption or surgery
* Those who have hypersensitivity reaction or clinically significant hypersensitivity reaction in the history of Investigational product

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-07-02 (Actual); Primary Completion 2019-08-10 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Cmax | 0, 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14h
  Maximum concentration of DWJ1421
AUClast | 0, 0.17, 0.33, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 14h
  Area under the drug concentration-time curve

CONTACTS AND LOCATIONS:
Locations (1):
- Bundang CHA Medical Center, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shin W, Yang AY, Yun H, Cho DY, Park KH, Shin H, Kim A. Bioequivalence of the pharmacokinetics between tofacitinib aspartate and tofacitinib citrate in healthy subjects. Transl Clin Pharmacol. 2020 Sep;28(3):160-167. doi: 10.12793/tcp.2020.28.e13. Epub 2020 Sep 21. PMID 33062629